CLINICAL TRIAL: NCT02218086
Title: Effectivity of Slackline-Training in Physiotherapy - a Randomised Controlled Study
Brief Title: Effectivity of Slackline-Training in Physiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: THIM - die internationale Hochschule für Physiotherapie (Other)
Collaborators: Vrije Universiteit Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UCP-2014-0107; KEK-ZH-2014-0107 (Registry Identifier: Kantonale Ethikkommission Zürich); PB 2019-00009 (Other: Kantonale Ethikkommission Zürich)
Record Dates: First submitted 2014-08-12; First posted 2014-08-15 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2019-05

CONDITIONS: Healthy Volunteers; Persons With no Known Significant Health Problems
Keywords: postural control; postural balance; slackline

STUDY DESIGN:
Intervention Model Description: different protocol-arms: crossover for comparing slackline vs. wobble board vs. flamingo balance task parallel for slackline training vs. enhanced standing-on-1-leg training
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- professionals (Experimental): balancing on the slackline / wobbling board 3 times by 30 seconds balancing on the slackline with a fix visual anchor / moving visual anchor 3 times by 30 seconds
  Interventions: Device: Slackline; Device: Wobbling Board; Device: Fix visual anchor; Device: Moving visual anchor
- beginners (Experimental): balancing on the slackline / wobbling board 3 times by 30 seconds pre-training compared to post-training
  Interventions: Device: Slackline; Device: Wobbling Board; Device: Pre-training; Device: Post-training; Device: Slackline vs. standing-on-1-leg vs. control

INTERVENTIONS:
Device: Slackline — Slackbase PRO CE: certificated by european law for medical devices (EG Richtlinie 93/42/EWG)
  Other Names: brand name: Slackbase PRO; http://medi-lines.com/slackbasepro/
Device: Wobbling Board — Wobbling Board CE: certificated by european law for medical devices (EG Richtlinie 93/42/EWG)
  Other Names: name: Standbrett; serial number: 2.1.1; http://www.originell.net/index.php?_disp=40
Device: Pre-training — First investigation of the beginners with less than 1 hour experience with slacklining.
  Arms: beginners
Device: Fix visual anchor — Professionals have to gaze at a fixed visual anchor during the slacklining.
  Arms: professionals
Device: Moving visual anchor — Professionals have to gaze at a moving visual anchor during the slacklining.
  Arms: professionals
Device: Post-training — Second investigation of the beginners occurs after a training session of 9 times 30 minutes within a few weeks.
  Arms: beginners
Device: Slackline vs. standing-on-1-leg vs. control — beginners have to train 9 times ~15minutes within y few weeks.
  Arms: beginners

SUMMARY:
Slacklines have been established in the last few years as a training equipment in sports such as climbing, skiing and others to increase postural control. Furthermore, slacklines are used in physiotherapy in terms of stabilizing training such as wobbling boards.

However, if slackline training is effective in rehabilitation has not been investigated yet. Therefore, to goal of this study will be to investigate the effectivity of slackline training in physiotherapy compared to a wobbling board with a single tilting axis.

Outcomes will be electromyographic-data and the kinetics of the whole body.

DETAILED DESCRIPTION:
Comparing beginners pre-training (less than 1 hour of slackline training) to post-training (9 times 30 minutes of individual, controlled training) to investigate the effects of balance training on a slackline.

Comparing beginners (less than 1 hour of slackline training) to professionals (more than 100 hours of slackline training) to investigate differences in balance strategies.

Comparing professionals during slacklining under two different conditions of their visual anchor: fix vs. moving. This to investigate the role of the visual system during balance reactions.

Comparing slackline training versus a demanding training standing-on-1-leg. We do compare Y-balance-performance, performance on the MFT challenge disc, each compared with simultanousely recording body Sway (lower trunk) with SwayStar.

Muscle activity will be investigated by absolute amplitude (mV) and frequency to get an idea of which muscle fibers are acting during the task and how the activation pattern may change through motor learning.

Body kinematics should show movement strategies especially differences in roll and pitch control of the body.

ELIGIBILITY:
Inclusion Criteria:

* young healthy, 18-30 years old
* small operations on muscle-skeletal-system on upper extremities
* birth control pill

Exclusion Criteria:

* any actual injuries on lower extremities
* injuries on lower extremities less than one year back
* operations of muscle-skeletal-system at shoulder/neck, trunk/pelvis and lower extremities
* fear of falling
* any medications
* cardiac pacemaker or cardiac arrhythmia
* pregnancy
* skeletal anomaly
* appendicitis less then 2 years back

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Muscle activity using surface electromyography device. 1. measuring amplitude of muscle activation in mV (millivolt) 2. measuring frequency pattern of muscle activation to distinguish /detect activation of slow and fast muscle fibers | average of 6 weeks
  single investigation for arms:
  1. BEGINNERS:
     a. slackline compared to wobble board
  2. PROFESIONALS:
     1. slackline compared to wobble board
     2. fix visual anchor compared to moving visual anchor
  double investigation: 1. BEGINNERS
  a. pre-training compared to post-training, expected training period average of 6 weeks, totally 9 trainings of 30 minutes each

SECONDARY OUTCOMES:
Whole body kinematics (composite outcome measure): a. calculating joint angles [deg & deg/s] b. calculating absolute and relative body part movements (such as trunk, pelvis, head): tilts & translations [mm, mm/s] | average of 6 weeks
  single investigation for arms:
  BEGINNERS:
  a. slackline compared to wobble board
  PROFESIONALS:
  slackline compared to wobble board fix visual anchor compared to moving visual anchor
  double investigation: 1. BEGINNERS
  a. pre-training compared to post-training, expected training period average of 6 weeks, totally 9 trainings of 30 minutes each

OTHER OUTCOMES:
measuring the duration of a trial (if less than 30 sec): measured in sec | average of 6 weeks
  single investigation for arms:
  BEGINNERS:
  a. slackline compared to wobble board
  PROFESIONALS:
  slackline compared to wobble board fix visual anchor compared to moving visual anchor
  double investigation: 1. BEGINNERS
  a. pre-training compared to post-training, expected training period average of 6 weeks, totally 9 trainings of 30 minutes each
Y-balance-performance: measured in cm | average of 6 weeks
  single investigation for arms:
  BEGINNERS:
  a. slackline training vs. standing-on-1-leg training vs. control
  a. pre-training compared to post-training, expected training period average of 6 weeks, totally 9 trainings of 15 minutes each
MFT challenge disc: measured in a score | average of 6 weeks
  single investigation for arms:
  BEGINNERS:
  a. slackline training vs. standing-on-1-leg training vs. control
  a. pre-training compared to post-training, expected training period average of 6 weeks, totally 9 trainings of 15 minutes each
  -------------------------------------- MFT Scale (Multi Functional Training)
  Scale Construct The diagnostics and scoring on the Challenge Disc is based on experience with other similar test equipment. Espacially the widely used Biodex Stability System.
  Total Score Total score is composed of the anterior-posterior and lateral-medial movement on the board.
  Scale Range Score 1-5 (1= good; 5=bad)
  Subscales unknown

CONTACTS AND LOCATIONS:
Overall Officials: Ursula M Kueng, PhD, Principal Investigator — THIM - die internationale Hochschule für Physiotherapie
Locations (1):
- Thim van der Laan University College Physiotherapy, Landquart, Kanton Graubünden, Switzerland

REFERENCES:
- [Background] Pfusterschmied J, Lindinger S, Buchecker M, Stoggl T, Wagner H, Muller E. Effect of instability training equipment on lower limb kinematics and muscle activity. Sportverletz Sportschaden. 2013 Mar;27(1):28-33. doi: 10.1055/s-0032-1330725. Epub 2013 Feb 12. PMID 23404457
- [Background] Donath L, Roth R, Rueegge A, Groppa M, Zahner L, Faude O. Effects of slackline training on balance, jump performance & muscle activity in young children. Int J Sports Med. 2013 Dec;34(12):1093-8. doi: 10.1055/s-0033-1337949. Epub 2013 May 22. PMID 23700328
- [Background] Honegger F, Tielkens RJ, Allum JH. Movement strategies and sensory reweighting in tandem stance: differences between trained tightrope walkers and untrained subjects. Neuroscience. 2013 Dec 19;254:285-300. doi: 10.1016/j.neuroscience.2013.09.041. Epub 2013 Oct 1. PMID 24090964
- [Background] Kung UM, Horlings CG, Honegger F, Duysens JE, Allum JH. Control of roll and pitch motion during multi-directional balance perturbations. Exp Brain Res. 2009 Apr;194(4):631-45. doi: 10.1007/s00221-009-1743-3. Epub 2009 Mar 5. PMID 19263044
- [Background] Raffi M, Piras A, Persiani M, Squatrito S. Importance of optic flow for postural stability of male and female young adults. Eur J Appl Physiol. 2014 Jan;114(1):71-83. doi: 10.1007/s00421-013-2750-4. Epub 2013 Oct 23. PMID 24150783
- [Background] Pfusterschmied J, Stoggl T, Buchecker M, Lindinger S, Wagner H, Muller E. Effects of 4-week slackline training on lower limb joint motion and muscle activation. J Sci Med Sport. 2013 Nov;16(6):562-6. doi: 10.1016/j.jsams.2012.12.006. Epub 2013 Jan 16. PMID 23333134
- [Background] Paoletti P, Mahadevan L. Balancing on tightropes and slacklines. J R Soc Interface. 2012 Sep 7;9(74):2097-108. doi: 10.1098/rsif.2012.0077. Epub 2012 Apr 18. PMID 22513724
- [Background] Kung UM, Horlings CG, Honegger F, Allum JH. The effect of voluntary lateral trunk bending on balance recovery following multi-directional stance perturbations. Exp Brain Res. 2010 May;202(4):851-65. doi: 10.1007/s00221-010-2201-y. Epub 2010 Mar 4. PMID 20204607
- [Background] Kung UM, Horlings CG, Honegger F, Allum JH. Incorporating voluntary unilateral knee flexion into balance corrections elicited by multi-directional perturbations to stance. Neuroscience. 2009 Sep 29;163(1):466-81. doi: 10.1016/j.neuroscience.2009.06.009. Epub 2009 Jun 6. PMID 19505537
- [Background] Tabira T, Sakai K. Demyelination induced by T cell lines and clones specific for myelin basic protein in mice. Lab Invest. 1987 May;56(5):518-25. PMID 2437389
- See also: Swiss National Clinical Trials Portal (SNCTP) — http://www.kofam.ch/